CLINICAL TRIAL: NCT00661882
Title: Integrated Cancer Repository for Cancer Research (iCaRe2)- Subproject: Pancreatic Cancer Collaborative Registry
Brief Title: Pancreatic Cancer Collaborative Registry
Status: Completed | Type: Observational
Sponsor: University of Nebraska (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 0405-02-FB; 5T32CA009476 (NIH)
Record Dates: First submitted 2008-04-18; First posted 2008-04-21 (Estimated); Last update posted 2023-09-06 (Actual); Status verified 2023-08

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; recurrent pancreatic cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Biopsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Questionnaire Blood: 30ml Access to leftover tissue: release a portion of leftover tissue collected and saved from surgery/biopsy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: medical chart review — Medical information, called "protected health information" (PHI), which includes demographic information (like address and birth date), the results of physical exams, blood tests, x-rays and other diagnostic and medical procedures and treatments, as well as medical and surgical history will be accessed from the subject's medical record.
Other: questionnaire administration — Provide or complete personal information about themselves, their medical history, their diet and lifestyle habits, any past or current environmental exposures and to re-create their family tree for any cancers that have occurred in any of their family members. In accordance with OPRR guidelines, no identifying information such as name, address, or date of birth will be used for relatives, but the affected status (cancer, age of onset, age of death) will be recorded. This information will be collected by whichever method they prefer; completing the questionnaires on hardcopy (to then be entered into the PCCR by a data manager) or by logging on to the PCCR website to complete the questionnaires by obtaining a user id and password to enter their information directly into the PCCR. Study participants who are in the EDRN project are required to complete the questionnaires on hardcopy (to then be entered into the PCCR by a data manager).
Other: study of socioeconomic and demographic variables — Share the information they provided with the PCCR research collaborators. This national group has formed the PCCR and is dedicated to pooling their efforts against pancreatic cancer.
Procedure: biopsy — Release a portion of pancreatic tissue, tumor tissue and/or metastatic pancreatic cancer tissue and/or paraffin embedded tissue that has already been collected and saved from their previous surgery or biopsy for storage in the UNMC Solid Tumor Bank for future studies done here or at collaborating institutions. All studies will be proposed in future IRB submissions.

SUMMARY:
RATIONALE: Gathering information about patients with cancer may help doctors learn more about the disease and plan early diagnosis and treatment.

PURPOSE: This clinical trial is studying computer tools for improving early diagnosis and treatment in patients with pancreatic cancer, are at risk for pancreatic cancer, or have a non-cancerous pancreatic disorder.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop Integrated Biomedical Computing Tools (IBCT) for the better understanding and treatment of pancreatic cancer by using the power of computer and informatics sciences.
* Continue development of the Pancreatic Cancer Collaborative Registry (PCCR) infrastructure to act as a repository for socio-demographic, environmental, clinical, and family history data collected from individuals and interested family members with a personal and/or family history of pancreatic cancer.
* Participate in an international pancreatic registry known as the PCCR by sharing information collected for research purposes only, to be used by pancreatic cancer research collaborators from other institutions.
* Collect and bank excess biological materials (i.e., pancreatic tissue, tumor tissue, and/or metastatic pancreatic cancer tissue, and/or paraffin-embedded tissue), blood, and serum from registry participants for future research.

OUTLINE: This is a multicenter study.

Patients undergo blood and pancreatic tissue collection. Normal, tumor, and/or metastatic pancreatic cancer tissue, and/or paraffin-embedded tissue from prior surgery or biopsy are obtained.

Patients provide or complete personal information about themselves, their medical history, their diet and lifestyle habits, any past or current environmental exposures, and re-create their family tree for any cancers that have occurred in any of their family members. Clinical data is collected annually.

High Risk participants provide blood samples and complete questionnaires at baseline. Clinical data is collected annually.

ELIGIBILITY:
Patients Participants Inclusion Criteria:

Must meet 1 of the following criteria:

* Histologically confirmed adenocarcinoma of the pancreas

  * Resectable stage I-IIA disease or stage IIB or higher disease Must have undergone complete surgical resection of the tumor with curative intent
  * Pancreatic mass (solid) that is less than 4 cm as determined by any conventional imaging (MRI, EUS, or CT scan)
  * No evidence of extension of the mass beyond the pancreas including vascular invasion or invasion into surrounding organs, with the exception of the bile duct
  * No imaging evidence of metastatic disease or lymphadenopathy (lymph nodes greater than 1 cm and/or appearance suspicious for an advanced lesion by imaging criteria)
* Has a family history of pancreatic cancer and is considered to be an at-risk individual for the disease (i.e., member of a family with 2 or more individuals with pancreatic cancer)

Patients Participants Exclusion Criteria:

* No prior malignancy, except nonmelanoma skin cancer, for 10 years
* No prior preoperative chemoradiotherapy (neoadjuvant)

Control participants Inclusion Criteria:

Must meet 1 of the following criteria:

* Chronic pancreatitis OR history of exocrine insufficiency meeting the following criteria:

  o At least 2 of the following criteria are met (unless patient has a history of pancreatic exocrine insufficiency in which case only 1 criterion must be met): Abdominal ultrasound that is consistent with chronic pancreatitis by standard radiological criteria (i.e., echogenic foci in the parenchyma, large or small cavities, calcifications, or dilated pancreatic duct) Abdominal CT scan consistent with chronic pancreatitis by standard radiological criteria (i.e., calcifications, dilated pancreatic duct, irregular contour of the gland, or cystic lesions) Endoscopic retrograde cholangiopancreatography exam consistent with chronic pancreatitis by standard radiological criteria (i.e., dilated tortuous main pancreatic duct with irregular secondary branches or intraductal calculi) Endoscopic ultrasound consistent with chronic pancreatitis by standard radiological criteria (i.e., echogenic foci, focal regions of decreased echogenicity, or pancreatic ductal changes)Pancreatic calcifications identified on plain film of the abdomen
* Must have an imaging study of the pancreas within 3 months of study enrollment that does not suggest a pancreatic mass
* Stable clinical history over the past year with no suspicion for cancer due to weight loss, jaundice, or change in abdominal symptoms
* Acute biliary obstruction (stones) including jaundice of benign etiology meeting the following criteria:
* Elevation of serum bilirubin level greater than 2.0 mg/dL
* Dilated extrahepatic biliary systems demonstrated on US, MRI, or CT scan
* Blood sample available within 72 hours of admission and prior to any corrective intervention
* Biliary obstruction must be of benign etiology such as common bile duct stone or benign biliary stricture
* Must have complete imaging study performed of the pancreas that does not suggest a pancreatic cancer (i.e., discrete mass lesion)
* Age, race, and sex-matched to qualified pancreatic cancer cases

Control Participants Exclusion Criteria:

* No family history of pancreatic cancer
* No personal history of acute pancreatitis or biliary obstruction (stones) including jaundice of benign etiology
* No concurrent abdominal pain
* No concurrent unexplained weight loss

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be asked to voluntarily participate in this project because they have been diagnosed with PC, have a family history of PC, or fulfill the criteria to be one of the three different control groups meaning they will either have a diagnosis of chronic pancreatitis, acute biliary obstruction, or they are a healthy unaffected individual.
Sampling Method: Non-Probability Sample
Enrollment: 379 (Actual)
Dates: Start 2003-02; Primary Completion 2013-09-09 (Actual); Study Completion 2013-09-09 (Actual)

PRIMARY OUTCOMES:
Development of the Pancreatic Cancer Collaborative Registry (PCCR) infrastructure as a repository for socio-demographic, environmental, clinical, and family history data | Yearly
  Ongoing registry.

CONTACTS AND LOCATIONS:
Overall Officials: Quan Ly, MD, Principal Investigator — University of Nebraska
Locations (1):
- Eppley Cancer Center, University of Nebraska Medical Center, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No